CLINICAL TRIAL: NCT00264732
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study of Amolimogene (ZYC101a) in the Treatment of High-Grade Cervical Intraepithelial Lesions (CIN 2/3) of the Uterine Cervix
Brief Title: A Study of Amolimogene (ZYC101a) in Patients With High Grade Cervical Intraepithelial Lesions of the Uterine Cervix
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYC1-004
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2012-05

CONDITIONS: Uterine Cervical Dysplasia
Keywords: cervical lesions; cervical dysplasia; Human papilloma virus; abnormal Pap; High-grade cervical intraepithelial lesions (CIN 2/3)
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — ZYC101a

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Amolimogene
- 2 (Experimental)
  Interventions: Drug: Amolimogene
- 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amolimogene — 1-dose amolimogene Group: Two intramuscular (IM) injections (100 micrograms ZYC101a per injection), one in each quadriceps, at Treatment Initiation. Single IM placebo injections (approximately 1 mL 0.9% sterile saline) at Weeks 3 and 6 in alternating quadriceps.
  Other Names: ZYC101a
  Arms: 1
Drug: Amolimogene — 3-dose amolimogene Group: Two IM injections (100 micrograms ZYC101a per injection), one in each quadriceps, at Treatment Initiation. Single IM injections of 100 micrograms ZYC101a at Weeks 3 and 6 in alternating quadriceps.
  Other Names: ZYC101a
  Arms: 2
Other: Placebo — Placebo Group: Two IM placebo injections at Treatment Initiation (1 injection in each quadriceps). Single placebo injections at Weeks 3 and 6 in alternating quadriceps. Each placebo injection consists of approximately 1 mL 0.9% sterile saline.
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of amolimogene, in the treatment of patients with high-grade cervical intraepithelial lesions of the uterine cervix.

DETAILED DESCRIPTION:
This is a double-blind study, so neither the patient not the doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be considered for enrollment, patients must:

1. Have an abnormal Pap smear (atypical squamous cells of undetermined significance [ASCUS], atypical squamous cells, cannot exclude high grade [ASC-H], low grade squamous intraepithelial lesion [LSIL], high grade squamous intraepithelial lesion [HSIL]) result within 6 months of screening visit.
2. Have a colposcopically visible lesion suspected to be high-grade that does not involve more than 75% of the cervix.
3. Have a CIN 2/3 consensus pathology diagnosis on tissue taken from a colposcopically-directed punch biopsy.
4. Not have evidence of cervical carcinoma on Pap smear or biopsy and not have a positive endocervical curettage.
5. Not have atypical endometrial cells or glandular-cell atypia on Pap smear or biopsy.
6. Have colposcopic visualization of entire squamocolumnar junction and of the entire lesion (i.e. cannot extend into canal).
7. Not have concomitant cancer, history of malignancies, including carcinoma of the cervix, except for non-melanoma skin cancer.
8. Be willing to sign an Institutional Review Board (IRB) approved informed consent. Minors must have the consent of a parent or legal guardian as required by local laws and regulations.
9. Agree to use 2 acceptable forms of contraception (e.g., double-method including at least one barrier and one hormonal method).
10. Be capable of complying with the protocol.
11. Not have other illnesses that would put the patient at undue risk for participation in the trial or would interfere with the required clinical observations.
12. Not have abnormalities of hematological, renal, or hepatic function as determined by clinical laboratory testing.
13. Not have immunologic disorder such as immunodeficiency, lupus, or other chronic auto-immune disease.
14. Not have an active systemic infection requiring treatment.
15. Not have ongoing systemic chronic steroid therapy or immunosuppressive medication (inhalers used for treating asthma and topical steroids are permitted).
16. Not be positive for HIV antibody.
17. Not be pregnant or lactating.
18. Not plan to use a cervical cap or diaphragm during the study.
19. Not have been treated with any investigational agent within 30 days prior to randomization in this trial.
20. Not have had prior gene therapy.
21. Not have had an excisional or ablative procedure performed on the cervix within one year of enrollment.
22. Be willing to consent to an excisional procedure, such as LEEP or cold-knife cone procedure, if indicated.

Please note: There may be additional inclusion/exclusion criteria. The study center will determine if patients meet all of the criteria. If patients do not qualify for the trial, study personnel will explain the reasons. If patients do qualify, study personnel will explain the trial in detail using an IRB-approved informed consent, and answer any questions. Patients can then decide if they wish to participate.

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 251 (Actual)
Dates: Start 2005-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Cervical intraepithelial neoplasia (CIN) 2/3 resolution, defined as the histological evaluation of cervical tissue (presence or absence of CIN 2/3 as determined by pathology consensus diagnosis) at the End of Observation (EOO) period. | 24 weeks after enrollment.

SECONDARY OUTCOMES:
Histology based on biopsy to determine the proportion of pts. w/resolution of CIN2/3. This is the same as primary efficacy variable in determination of presence or absence of CIN2/3, but excludes pts. with excisional procedure or cytology information. | 24 weeks after enrollment.
Histological resolution to normal to examine the proportion of patients with a histology result of "normal" versus "abnormal." | 24 weeks after enrollment.
Clearing or persistence of lesions based on colposcopic findings to examine the proportion of patients with "no lesion" versus "at least one lesion." | 24 weeks after enrollment.
Pap smear cytology. | 24 weeks after enrollment.
Clearing or persistence of original human papillomavirus (HPV) subtype as determined by HPV typing to present the number and percent of patients with absence of all HPV. | 24 weeks after enrollment.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of Alabama, Birmingham, Alabama
  - Arizona Wellness Center for Women/Precision Trials, LLC, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Arrowhead Regional Medical Center, Colton, California
  - The Center for Advanced Research and Education, Inc., Palm Springs, California
  - Medical Center for Clinical Research, San Diego, California
  - Physicians Research Options, LC, Lakewood, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - University of Florida, Miami, Miami, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Insignia Clinical Research, Tampa, Florida
  - Comprehensive Clinical Trials LLC, West Palm Beach, Florida
  - Medical College of Georgia, Department of Family Medicine, Augusta, Georgia
  - Rosemark Women's Care Specialists, Idaho Falls, Idaho
  - University of Minnesota, Minneapolis, Minnesota
  - Centennial Hills OB-GYN Associaties, North Las Vegas, Nevada
  - Southwest Clinical Research, Albuquerque, New Mexico
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - The University of Oklahoma Health Sciences Center, Center for Research in Women's Health, Oklahoma City, Oklahoma
  - Temple Center for Women's Health, Philadelphia, Pennsylvania
  - Sarah Cannon Research, Memphis, Tennessee
  - Michael Altenbern, MD, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Physicians' Research Options, Pleasant Grove, Utah
  - Physicians' Research Options, LLC, Sandy City, Utah
  - Tidewater Clinical Research, Virginia Beach, Virginia

REFERENCES:
- [Background] Crum CP, Beach KJ, Hedley ML, Yuan L, Lee KR, Wright TC, Urban RG. Dynamics of human papillomavirus infection between biopsy and excision of cervical intraepithelial neoplasia: results from the ZYC101a protocol. J Infect Dis. 2004 Apr 15;189(8):1348-54. doi: 10.1086/382956. Epub 2004 Mar 30. PMID 15073670
- [Background] Garcia F, Petry KU, Muderspach L, Gold MA, Braly P, Crum CP, Magill M, Silverman M, Urban RG, Hedley ML, Beach KJ. ZYC101a for treatment of high-grade cervical intraepithelial neoplasia: a randomized controlled trial. Obstet Gynecol. 2004 Feb;103(2):317-26. doi: 10.1097/01.AOG.0000110246.93627.17. PMID 14754702